CLINICAL TRIAL: NCT01644058
Title: Immediate Loading Of Dental Implants In Mandible Full-Arch: A Pilot Clinical Study On Patients Satisfaction, Quality Of Life And Implant Success
Brief Title: Immediate Loading Of Dental Implants: A Pilot Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Elham Emami, D.D.S., M. Sc., Ph. D, Professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDEM-EE-2012b
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Dental Implantation
Keywords: immediate-loading; patient-based outcomes
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Masking Description: Investigators were not involved in data analysis
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immediate loading (Experimental): Immediate loading of 2 endo-osseous mandibular implants
  Interventions: Procedure: Immediate loading

INTERVENTIONS:
Procedure: Immediate loading
  Other Names: Procedure: Immediate loading of 2 endo-osseous unsplinted implants of a mandibular overdenture

SUMMARY:
Objective: To provide 2-year clinical- and patient-oriented data with regard to mandibular overdenture assisted by 2 immediately loaded unsplinted implants.

DETAILED DESCRIPTION:
In this pre-post design, Phase-I clinical trial, 18 edentate individuals received a new set of complete denture. Then, following standard procedures, 3 threaded implants (OsseoSpeed TXTM, Dentsply Implants, Mölndal, Sweden) were placed in the mandible in each patient, and locator abutments (Zest Anchors LLC, Escondido, U.S.A.) were inserted on the right and left side implants. The midline implant served as a control for within-patient comparison. The immediate loading was conducted within 24 h of surgery. Data were collected at baseline (T0), 12 (T1) and 24 (T2) months after immediate loading. The clinical outcomes included implant survival rate, crestal bone level changes and implant stability. These criteria were assessed through clinical and radiographic examinations as well as resonance frequency analysis. Patient-centered outcomes included patient satisfaction and oral health-related quality of life measured using validated questionnaires. Brunner-Langer approach was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age of 18 years
* Complete edentulism for more than 1 year
* Wear of total conventional prosthesis for more than 1 year
* Bone morphology in the anterior mandibular region amendable for the placement of 3 regular diameter implants without any additional procedure (graft or membrane).

Exclusion Criteria:

* Any absolute or relative contra-indication to implant therapy
* Physical incapacity to render oral or prosthetic hygiene
* Incapacity to obtain a free and informed consent
* Incapacity to assist to planned follow up appointments
* Incapacity to understand and complete questionnaires

Exclusion Criteria to Immediate Loading Protocol Found on One or Both of Un-splinted Implants During Surgery:

* Inadequate bone quality: IT<35 Ncm
* Inadequate primary stability: ISQ<60

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elham Emami, DDS, MSc,PhD, Principal Investigator — Université de Montréal, Faculty of Dentistry
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Calling patients on the waiting list of the undergraduate implant clinic of the Université de Montréal and referrals from active study subjects.
Period: Overall Study
Arm/Group | Immediate Loading
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Immediate Loading
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Region of Enrollment [Number; unit: participants]
  Canada | 18

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With the Immediate Loading Protocol
Description: Visual Analogue Scale (VAS) to assess patients' satisfaction, with a score of 100 being extremely satisfied (minimum and maximum scores: 1-100 respectively).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Immediate Loading
Number analyzed (Participants) | 18
millimeters | 40.3 (34.9) [0 to 99]

2. Primary Outcome: Oral-health-related Quality of Life With the Immediate Loading Protocol
Description: Oral Health Impact Profile (OHIP-20) to assess oral-health-related quality of life: score ranges between 20 and 120 points, with a lower score indicating a better oral-health-related quality of life.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Immediate Loading: Immediate loading of 2 endo-osseous mandibular implants
  Immediate loading
Arm/Group | Immediate Loading
Number analyzed (Participants) | 18
units on a scale | 66.8 (19.1)

ADVERSE EVENTS:
Time Frame: All participants were assessed for adverse events. "0" participants were found to have serious or non-serious events after observation.
Arm/Group | Immediate Loading
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
Phase-I clinical trial with small sample size and a pre-post design with no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes